CLINICAL TRIAL: NCT06278493
Title: A Phase I/IIa Clinical Trial AL2846 Capsule Combined With Gemzar Injection in the Treatment of Advanced Pancreatic Cancer.
Brief Title: A Clinical Study of AL2846 Capsule Combined With Gemzar Injection in the Treatment of Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL2846-I-0002
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AL2846 capsules + Gemzar injection (Experimental): AL2846 capsules combined with Gemzar injection,28 days as a treatment cycle
  Interventions: Drug: AL2846 capsules; Drug: Gemzar

INTERVENTIONS:
Drug: AL2846 capsules — AL2846 is a multi -target receptor tyrosine kinase inhibitor.
Drug: Gemzar — It is a chemotherapeutic drug.

SUMMARY:
This is a clinical study to observe the tolerance and primary efficacy of AL2846 capsules combined with Gemzar injection in patients with pancreatic cancer, and to determine the recommended dosage and administration method for subsequent clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Non operative patients with pancreatic cancer confirmed by histology or cytology, At least one evaluable lesion exists.
* ≥18 years old and ≤70 years old, Eastern Cooperative Oncology Group (ECOG) Performance Status: 0-1, expected survival period of more than 3 months.
* No chemotherapy or targeted treatment has been carried out for advanced pancreatic cancer, or more than half a year after the end of postoperative treatment.
* Normal function of major organs.
* Female subjects should agree to use contraception during the study period and within 6 months after the end of the study; Within 7 days prior to enrollment in the study, the serum or urine pregnancy test should be negative and must be a non lactating patient; Male subjects should agree to use contraceptive measures during the study period and within 6 months after the end of the study period.
* Subjects voluntarily participate in this study and sign informed consent.

Exclusion Criteria:

* Have any type of active malignant tumor or have a history of malignant tumor.
* Previously treated with Gemzar injection.
* Known brain metastases, spinal cord compression, cancerous meningitis, or diseases of the brain or pia mater detected during Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) screening.
* Clinically significant ascites in patients.
* Diarrhea greater than or equal to level 2.
* Have any acute or chronic active infectious disease.
* Hypertensive patients who cannot be well controlled, or suffering from myocardial ischemia or myocardial infarction, arrhythmia, and grade I heart failure.
* Urine routine indicates urine protein ≥++, and it is confirmed that the 24-hour urine protein quantification is greater than 1.0 g.
* History of abdominal fistula, gastrointestinal perforation, or abdominal abscess within 6 months.
* Long term unhealed wounds or fractures.
* Individuals who have experienced arterial/venous thrombosis events within 6 months, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis, and pulmonary embolism.
* Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or their analogues; Under the premise that international normalized ratio (INR) is ≤ 1.5, it is allowed to use low-dose warfarin (1mg orally, once daily) or low-dose aspirin (not exceeding 100mg daily) for preventive purposes.
* Individuals with a history of psychiatric drug abuse who are unable to quit or have mental disorders.
* Patients known to be allergic to Gemzar injection.
* Patients with active hepatitis B or hepatitis C.
* Individuals with a history of immunodeficiency, including HIV testing positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
* According to the investigator's judgment, there are accompanying diseases that seriously endanger patient safety or affect the completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Up to 4 weeks.
  One or more unacceptable toxic reactions that appear after administration cause the dose or extend the dose cycle that cannot continue to increase the dose or extend the dose
Maximum tolerated dose (MTD) | Up to 4 weeks.
  If dose limiting toxicity (DLT) occurs in 2 or more subjects in a given dose group, the dose level in the previous dose group is considered MTD.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China